CLINICAL TRIAL: NCT05042518
Title: The Effectiveness of Psychological Skill Training on Quantitative Electroencephalogram (EEG) in Athletes Before the Competition
Brief Title: Psychological Skill Training for Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: ANanbancha
Record Dates: First submitted 2021-09-01; First posted 2021-09-13 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: No Conditions

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The participant in the intervention group will practice breathing control and self-talk with objectives for relaxation. The duration of training is 4-5 minutes in each session, 4 sessions per week for 1 month.
  Interventions: Behavioral: Experiment
- Control group (Placebo Comparator): The participant in the control group will receive consultations by a sport psychologist for goal setting and positive thinking. The duration is similar to the training group (4-5 minutes in each session, 4 sessions per week for 1 month).
  Interventions: Other: Control

INTERVENTIONS:
Behavioral: Experiment — breathing control and self-talk with objectives
  Arms: Intervention group
Other: Control — The participant in the control group will receive consultations by a sport psychologist for goal setting and positive thinking. The duration is similar to the training group (4-5 minutes in each session, 4 sessions per week for 1 month)
  Arms: Control group

SUMMARY:
The investigator will determine the effectiveness of psychological skill training on quantitative EEG in athletes before the competition.

DETAILED DESCRIPTION:
Psychological skills training is the mental training that can apply for increased athletes' performance to make athletes more confident. The objective of psychological skill training is to develop the potential of athletes to be able to show their abilities (Peak Performance), and to create satisfaction, self-esteem, for athletes. Additionally, the ability to concentrate and reduce anxiety could affect athletes' emotions and be ready to participate in the competition. Therefore, this study will apply psychological skills training for athletes. The effectiveness of psychological skill training will be measured by using quantitative EEG before and after training. The quantitative EEG assessments could demonstrate an anxiety level at different stages of the competition and it could reveal the changes caused by training. The intervention will begin 3 months before the competition. The quantitative EEG measurements are arranged 4-5 times following the previous study. The sequence of the measurement will be including a baseline: one month before the competition, two weeks before the competition, a week before the match, three days before the match (depend on the situation), three days after the match (post-training).

ELIGIBILITY:
Inclusion Criteria:

* Athletes male or female
* Age between 18-35

Exclusion Criteria:

* Having an acute injury to the musculoskeletal structures of other joints of the lower extremity in the previous 3 months

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2022-04-05 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
ฺBrain wave | Through study completion, an average of 5 weeks
  to identify psychological change

SECONDARY OUTCOMES:
Revised Competitive State Anxiety Inventory: CSAI - 2R | Through study completion, an average of 5 weeks
  Questionnaire for evaluate anxiety level. The participants will circle the number on the Likert scale from 1 to 4 of how they feel in that moment. The numbers 1 to 4 represent the following statements : 1 = Not at all 2 = Somewhat 3 = Moderately so 4 = Very much so. A higher score presents a higher anxiety level.

CONTACTS AND LOCATIONS:
Overall Officials: Kittichai Tharawadeepimuk, Dr, Principal Investigator — College of sports science and technology, Mahidol University, Thailand
Locations (1):
- Mahidol University, Salaya, Nakhonprathom, Thailand

IPD SHARING:
Plan to Share IPD: No